CLINICAL TRIAL: NCT02071069
Title: Efficacy and Tolerance of Cetuximab Combined With Irinotecan or Fluorouracil as Maintenance Therapy in Patients With RAS-wild-type Incurable Advanced Colorectal Cancer （Confirm Study）
Brief Title: Efficacy and Tolerance of Maintenance Therapy in Patients With Incurable Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianshu Liu (Other)
Responsible Party: Sponsor-Investigator, Tianshu Liu, Director of Medicine-Oncology department, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-ON-05
Record Dates: First submitted 2014-02-19; First posted 2014-02-25 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Incurable Colorectal Cancer; RAS-wild-type
Keywords: Incurable colorectal cancer; maintenance therapy; Cetuximab
MeSH Terms: interventions — Cetuximab; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- maintenance therapy (Experimental): Initially, all subjects received 8 cycles of Cetuximab (400mg/m2 d1,250mg/m2 every week or 500mg/m2 every 2 weeks)plus FOLFIRI (irinotecan 180 mg/m2 IV on day 1 , leucovorin 400mg/m2 on day 1 , fluorouracil 400mg/m2 on day 1 and fluorouracil 2400mg/m2 civ46h every 2 weeks) .
  After 8 cycles or severe toxicity, patients received maintenance therapy comprising Cetuximab (250mg/m2 every week or 500mg/m2 every 2 weeks) and either irinotecan( 180 mg/m2 IV every 2 weeks) or fluorouracil arm( leucovorin 400mg/m2 on day 1 , fluorouracil 400mg/m2 on day 1 and fluorouracil 2400mg/m2 civ46h every 2 weeks ). In cases of unacceptable toxicity, only the related medication was stopped
  Interventions: Drug: Cetuximab; Drug: irinotecan; Drug: fluorouracil

INTERVENTIONS:
Drug: Cetuximab — 400mg/m2 d1,250mg/m2 every week or 500mg/m2 every 2 weeks
Drug: irinotecan — 180 mg/m2 IV every 2 weeks
Drug: fluorouracil — 400mg/m2 on day 1 and 2400mg/m2 civ46h every 2 weeks
  Other Names: 5FU

SUMMARY:
1. To evaluate efficacy, safety, and feasibility of maintenance therapy with Cetuximab combined with irinotecan or fluorouracil after Cetuximab plus irinotecan and fluorouracil(FOLFIRI) in patients with incurable colorectal cancer.
2. The relevant phase III studies reported that the progression free-survival of cetuximab combined with FOLFIRI in advanced colorectal cancer was 4.3 months up to 6.8 months.

This study assumed that the progression free-survival was 5.1 months which was not inferior to the continuous chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years with histologically confirmed metastatic colorectal cancer
2. Eastern Cooperative Oncology Group performance status ≤2 and
3. life expectancy of >3 months were enrolled.
4. All patients had to have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1)
5. None was previous exposure to Cetuximab or irinotecan .
6. Patients had to have adequate haematological (absolute neutrophil count >1.5 × 109/l; platelet count >100 × 109/l; haemoglobin >9 g/dl), hepatic [total bilirubin <1.5 × the upper limit of normal (ULN); alanine aminotransferase and aspartate aminotransferase <2.5 × ULN, or <5 × ULN in the case of hepatic metastases or <10 × ULN in the case of osseous metastases; alkaline phosphatase <2.5 × ULN, or <5 × ULN or <10 × ULN in the case of hepatic or osseous metastases, respectively] and renal function (creatinine clearance ≥60 ml/min)
7. All RAS were wildtype. -

Exclusion Criteria:

1. Pregnant or breast-feeding women;
2. Clinically significant cardiac disease;
3. Lack of physical integrity of the upper gastrointestinal tract;
4. History of other malignancy;
5. Central nervous system metastases. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The progression free-survival | 8 Months after the last subject participate in
  defined as the time from enrollment to progression or death RECIST guidelines were used to define all responses after patients had received every 8 weeks of therapy

SECONDARY OUTCOMES:
Overall survival | 18 Months after the last subject participate in
  defined as the time from enrollment to death
Grade 3 and 4 adverse Events as a Measure of Safety and Tolerability | 3 Months after the last subject end the treatment
  Toxicity was graded according to the criteria of the National Cancer Institute Common Terminology for Adverse Events (version 4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, Doctor, Principal Investigator — Medicine-Oncology Derpartment of Zhongshan hospital
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China